CLINICAL TRIAL: NCT00300560
Title: Efficacy and Safety of Colistin for Therapy of Infections Caused by Extended Spectrum Beta-Lactamase(ESBL) Producing Klebsiella Pneumoniae or Escherichia Coli
Brief Title: Efficacy and Safety of Colistin for Therapy of Infections Caused by ESBL Producing K.Pneumoniae or E.Coli
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SirirajCEU49-004
Record Dates: First submitted 2006-03-07; First posted 2006-03-09 (Estimated); Last update posted 2006-05-22 (Estimated); Status verified 2006-03

CONDITIONS: Infections
Keywords: ESBL-producing E.coli Infections; ESBL-producing Klebsiella pneumoniae Infections; Colistin
MeSH Terms: conditions — Infections | interventions — Colistin

INTERVENTIONS:
Drug: Colistin

SUMMARY:
In patients with documented ESBL-producing E.coli and Klebsiella pneumoniae will be allocated to receive colistin or conventional antibiotic regimen.

DETAILED DESCRIPTION:
In patients with documented ESBL-producing E.coli and Klebsiella pneumoniae will be allocated to receive colistin or conventional antibiotic regimen.The primary outcome is clinical response and secondary outcomes are microbiological response and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 yr.
* Hospitalized to Siriraj Hospital
* Infections with ESBL-producing E.coli or K.pneumoniae
* Consent informed consent

Exclusion Criteria:

* Pregnancy or lactating mother
* Colistin allergy
* Neurologic diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152
Dates: Start 2006-02; Study Completion 2006-12

PRIMARY OUTCOMES:
Clinical response

SECONDARY OUTCOMES:
Microbiological response

CONTACTS AND LOCATIONS:
Overall Officials: Visanu Thamlikitkul, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Division of Infectious disease and Tropical Medicine, Department of Medicine, Faculty of Medicine Siriraj Hospital, Bangkoknoi, Bangkok, Thailand